CLINICAL TRIAL: NCT01058369
Title: Early Treatment With Deferasirox (Exjade®) in Low Risk MDS - a Prospective Multicentre Single-arm Single-stage Phase II Study -
Brief Title: Exjade-Early-Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient patient recruitment (only 2 patients)
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CICL670ADE06T
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Results first posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Deferasirox

ARMS (1):
- Deferasirox (Experimental)
  Interventions: Drug: Deferasirox (Novartis Pharma)

INTERVENTIONS:
Drug: Deferasirox (Novartis Pharma) — Treatment period 102 weeks. Starting dose 10mg/kg/day. Up to 30/mg/kg according to dose adjustment table as specified in the protocol
  Other Names: Exjade(R)

SUMMARY:
Study outline: Deferasirox (Exjade®) is regularly used in severe iron overload in order to avoid organ damage of liver, heart and other organs. It has been proposed, that iron overload may not only impose damage to other organs but also to the bone marrow and thus worsen hematopoietic insufficiency in patients with MDS. Patients presenting with low or INT-1 risk MDS with only mild iron overload will be treated with deferasirox in this study. It will be analyzed if hematological improvement can be observed during this treatment.

ELIGIBILITY:
Inclusion Criteria:

* MDS of subtype RA, RARS, RCMD, RCMD-RS (i.e. lower risk)
* RAEB I allowed, if clinically stable for > 3 months
* 5q-minus syndrome allowed, if lenalidomide unsuccessful or unavailable at the time of inclusion
* IPSS score < intermediate-1
* transfusion dependent or Hb < 10,5 g/dl
* History of less than 20 units of red blood cell transfusions or 100mL/kg of prepacked red blood cells (PRBCs), except for transfusions for acute bleeding
* Serum ferritin > 300 µg/l and < 1500 μg/l. This level should have been verified at least at two occasions within 3 months. Samples must be obtained in the absence of concomitant severe infection
* no indication for EPO (due to high endogenous EPO levels) or EPO without benefit in the past
* no indication and/or no plans for cytostatic drugs
* no previous exposure to cytostatic drugs, thalidomide, lenalidomide, G-CSF or EPO or exposure to any of these drugs has been terminated since > 8 weeks (4 weeks for G-CSF).
* no indication and/or no plans for stem cell transplantation
* stable or worsening cytopenia during the past 8 weeks. If in doubt, extend screening period to >= 8 weeks
* Patients of either gender and age > 18 years
* Life expectancy > 12 months
* Females of childbearing potential must use double-barrier contraception (for example orale contraception and condom).
* Mental ability of the patient to understand explications concerning the study and to understand and follow instructions of the investigating physician
* Written informed consent by the patient

Exclusion Criteria:

* Treatment with deferasirox or other chelation therapy for periods > 4 weeks before study start
* Patients with intolerance to Deferasirox
* Patients with a concomitant second malignant disease, possibly interfering with life expectancy
* Patients with mean levels of alanine aminotransferase (ALT) > 5x ULN
* Patients with uncontrolled systemic hypertension
* Patients with serum creatinine > 1.5x the upper limit of normal (ULN) or a creatinine clearance < 60 ml/min according to the MDRD formula (Levey 2005)
* History of nephrotic syndrome
* Systemic diseases (cardiovascular, renal, hepatic, etc.) which would prevent the patient from undergoing study treatment
* Patients with psychiatric or addictive disorders which prevent them from giving their informed consent or undergoing study treatment
* Patients treated with systemic investigational drugs within the past 4 weeks or topical investigational drug within the past 7 days
* Any other surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug. The investigator should be guided by evidence of any of the following:
* history of inflammatory bowel syndrome, gastritis, ulcers, gastrointestinal or rectal bleeding;
* history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection;
* history of pancreatic injury or pancreatitis; indications of impaired pancreatic function/injury as indicated by abnormal lipase or amylase;
* history of urinary obstruction or difficulty in voiding
* History of non-compliance to medical regimens and patients who are considered potentially unreliable and/or not cooperative
* History of drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by laboratory assays conducted during the screening period
* Patients with active uncontrolled infectious disease
* Pregnancy or breast feeding
* QT > 470 msec on screening ECG
* Patients with a history of Torsades de Pointes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Krause, Prof. Dr., Study Chair — Medizinische Klinik 5, Universitätsklinikum Erlangen
Locations (1):
- Medizinische Klinik 5, Universitätsklinikum Erlangen, Erlangen, Bavaria, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Deferasirox
Started | 2
Completed | 0
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Early termination study | 1

BASELINE CHARACTERISTICS:
Arm/Group | Deferasirox
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 42.5 [40 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  Germany | 2

OUTCOME MEASURES:

1. Primary Outcome: Fraction of Patients With Hematologic Improvement According to Modified IWG Criteria (Reduction of Transfusions and/or Increase in Hb, Improvement of Neutropenia and Thrombocytopenia)
Time Frame: within two years
Population: Trial prematurely ended due to insufficient recruitment before Primary endpoint was reached by any subject
Arm/Group | Deferasirox
Number analyzed (Participants) | 0

2. Secondary Outcome: Evaluate the Safety and Tolerability Profile of Deferasirox in MDS Patients
Time Frame: within two years
Reporting Status: Not Posted

3. Secondary Outcome: Effectiveness of Iron Depletion
Time Frame: within two years
Reporting Status: Not Posted

4. Secondary Outcome: Correlation Between Hematological Improvement and Effectiveness of Iron Depletion
Time Frame: two years
Reporting Status: Not Posted

5. Secondary Outcome: Development of Bone Marrow Morphology
Time Frame: two years
Reporting Status: Not Posted

6. Secondary Outcome: Correlation Between Hematological Improvement and Pretreatment Parameters. Extension of This Analysis to MDS Patients on Deferasirox Within the Licensed Indication (More Severe Iron Overload)
Time Frame: two years
Reporting Status: Not Posted

7. Secondary Outcome: Overall Survival
Time Frame: within two years
Reporting Status: Not Posted

8. Secondary Outcome: AML-free Survival
Time Frame: within two years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Deferasirox
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferasirox (N=2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
acute myeloid leukaemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferasirox (N=2)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
haematoma (Vascular disorders) | 1 (1)
thrombophlebitis (Vascular disorders) | 1 (1)
fatigue (General disorders) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
depression (Psychiatric disorders) | 1 (1)
wound (Injury, poisoning and procedural complications) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 1 (1)
abdominal pain upper (Gastrointestinal disorders) | 1 (1)
hypertension (Vascular disorders) | 1 (1)
emotional distress (Psychiatric disorders) | 1 (1)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
gingival bleeding (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early Termination leading to small numbers of subjects enrolled; number of subjects analysed = 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes